CLINICAL TRIAL: NCT05566327
Title: De-implementing Wisely: Using a Theory-based De-implementation Intervention to Reduce Low-value Preoperative Testing in Alberta
Brief Title: De-implementing Low Value Preoperative Care Wisely
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: The Ottawa Hospital (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-1173
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-09

CONDITIONS: Surgery-Complications; Anesthesia Complication
Keywords: Low value preoperative testing; Choosing Wisely CAnada

STUDY DESIGN:
Intervention Model Description: Randomized intervention trial
Who Masked: Outcomes Assessor
Masking Description: This is a health services intervention so the intervention and control group will know their allocation. The study team will know the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Clinics in this arm will receive the usual information about low value preoperative testing. Staff at these hospitals may be aware of the Choosing Wisely Anaesthesia Guidelines for reducing unnecessary testing, the Ontario Anaesthesiology Toolkit to operationalize the Choosing Wisely guidelines.
- Intervention Group (Active Comparator): The intervention will focus on increasing accountability for preoperative test ordering to reduce the number of inappropriate tests ordered for patients having ambulatory surgeries. A multi-component approach will be used to address the accountability of who should order preoperative tests for patients undergoing ambulatory surgery.
  Interventions: Behavioral: De-implementation Bundle

INTERVENTIONS:
Behavioral: De-implementation Bundle — A multicomponent intervention directed at the drivers of low value preoperative testing.
  An administrative change will be implemented whereby medically necessary preoperative tests for patients undergoing scheduled surgery will be ordered at the discretion of a consulting anaesthesiologist only. Workshops will be delivered to surgical, internal medicine, and anaesthesia divisions. The workshop program will include rationale for the policy, discussion of perceived local barriers to implementation and mitigation strategies.The clinical departments will commit to supporting the change in policy. Nurses will be coached to feel comfortable calling the anesthesiologist about any preoperative tests ordered, and the PAC nurses will have the authority to cancel tests. Check boxes will be removed from surgeons' and family physicians' order forms to reduce to ease of ordering the tests.
  Arms: Intervention Group

SUMMARY:
Low value preoperative testing does not improve patient outcomes or reduce adverse events. Low value preoperative testing costs patients and healthcare systems without benefit. In a previous study, the investigators identified the systems-level and individual-level drivers of low value preoperative testing.

In this study, the investigators will use these drivers of low value testing to design and implement a bundled intervention to reduce low value preoperative testing in Alberta, Canada. The investigators will measure the impact of this intervention on the number of low value tests, adverse events (ICU admissions, length of stay, 30-day readmissions), and patient costs. The investigators will also interview healthcare providers on their experiences with the intervention.

DETAILED DESCRIPTION:
Low-value care is defined as a test or treatment for which there is no evidence of patient benefit or where there is evidence of more harm than benefit. Choosing Wisely Canada (CWC) is a professionally led campaign that rallies medical professional to address the issue of low value care. For example, the CWC anaesthesiology recommendations produced by the Canadian Anaesthesiologists' Society recommends against baseline ordering of pre-operative tests.

Whilst the identification of potential areas of low-value care is an important first step in addressing this problem, the issue of implementing Choosing Wisely (CW) like recommendations has not received adequate attention

In the investigators previous study based on the Theoretical Domains Framework (TDF) (REB18-1097), they identified the factors that influence test ordering before low-risk surgical procedures. Barriers identified included conflict about who was responsible for the test-ordering (Social/professional role and identity), inability to cancel tests ordered by fellow physicians (Beliefs about capabilities and Social influences), and logistic problems with tests being completed before the anesthesiologists see the patient (Beliefs about capabilities and Environmental context and resources). There were also concerns that not testing might be associated with harms (Beliefs about Consequences). These findings led to the development of a theory-informed intervention that identifies anesthesiologists as primarily responsible for ordering of tests and strengthens accountability within hospitals. The next phase involves evaluating the theory-informed intervention.

The investigators will conduct a cluster randomized controlled trial in 20 hospitals in Alberta, Canada to evaluate whether the theory-based intervention to improve accountability can decrease the use of low-value tests before non-urgent surgery in otherwise healthy patients

Objectives The overall aim of this trial is to evaluate whether a theory-based intervention that addresses barriers and facilitators of persistent low value test ordering reduces low-value preoperative test (ECGs and CXRs) in patients undergoing low risk surgery.

The specific objectives are to:

1. Evaluate whether the intervention leads to a decrease in low-value preoperative test ordering compared to the control arm (standard of care).
2. Conduct a process evaluation to determine whether the intervention is delivered as designed (fidelity); to determine whether any changes in low-value preoperative test ordering are mediated through changes to the perceived barriers/enablers (mechanism of action); and to understand healthcare workers and patients experiences of the intervention.
3. Evaluate whether the intervention offers good value for money from the perspective of Canada's publicly funded health care system.

METHODS This pragmatic parallel arm cluster randomized controlled trial with pre- and post-intervention measurements will be conducted in hospitals that perform preoperative assessments (preadmission clinics, PACs) in Alberta, Canada. The intervention will be delivered to anaesthesiologists, surgeons, internists, pre-admission clinic nurses, and administrative staff responsible for the care for patients who are over 18 years of age and undergoing low-risk surgical procedures, defined as procedures with less than 1% mortality or cardiac events, including but not limited to endoscopy, ophthalmologic surgery, knee arthroscopy, hernia repair.

OBJECTIVE 1 Interventions Eligible hospitals will be randomly allocated to the intervention (multi-component intervention) and control arm (standard of care).

Intervention description The intervention will focus on increasing accountability for preoperative test ordering to reduce the number of inappropriate tests ordered for patients having ambulatory surgeries. A multi-component approach will be used to address the accountability of who should order preoperative tests for patients undergoing ambulatory surgery.

* Changing PAC and Hospital Policies
* Identification of a Local Champion
* Delivering an Education Workshop
* Restructuring Patient Flow and Responsibility

OBJECTIVE 2 The investigators will conduct a mixed-methods theory-based process evaluation alongside the trial. The evaluation will be performed through mechanistic sub-study (to determine whether our interventions activated the hypothesized mediating pathways and if so, was this sufficient to lead to implementation) and fidelity evaluation (to understand participants' experiences of being in a trial, and to determine whether the content of interventions was delivered as designed).

OBJECTIVE 3 The investigators will conduct a cost-effectiveness analysis from the perspective of Alberta Health. The total costs will include the costs of the intervention and observed harms associated with preoperative assessment (hospital admissions and re-operations).

ELIGIBILITY:
Inclusion Criteria:

* Low risk patient (no cancer, diabetes, or life-limiting disease)
* Undergoing a low-risk surgical procedure (a day surgery or any procedure with a less than 1% 30-day cardiac event or all-cause mortality)
* Adults
* Hospitals in the 26-100th centiles for low value preoperative test ordering

Exclusion Criteria:

* Has a life-limiting condition
* Pregnancy
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Low value preoperative testing | 1 year
  The proportion of patients undergoing one or more low value preoperative test (ECG, echocardiogram, chest x-ray or cardiac stress test) within 60-days of surgery

SECONDARY OUTCOMES:
Overnight admission | 1 year
  Proportion of patients who are admitted overnight to the hospital after low-risk surgery
Re-operation | 1 year
  Proportion of patients who require a second procedure during their hospital admission
ED Visits | 1 year
  Proportion of patients who represent to the emergency department within 30 days of their surgical discharge
Readmissions | 1 year
  Proportion of patients who are readmitted to hospital within 30-days of their surgery
ICU Admission | 1 year
  Proportion of patients who are admitted to an intensive care unit during their hospital admission
Length of stay | 1 year
  The length of stay for the surgical admission
Mortality | 1 year
  The proportion of patients who die from any cause within 30-days of their surgery

IPD SHARING:
Plan to Share IPD: Undecided
To be determined